CLINICAL TRIAL: NCT03570060
Title: Stepwise Screening for Silent Atrial Fibrillation After Stroke
Acronym: SAFAS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GUENANCIA 2017
Record Dates: First submitted 2018-06-07; First posted 2018-06-26 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sample — 2 ml of blood for testing for serum biomarkers (IL-6, GDF-15, soluble ST-2 soluble, osteoprotegerin, galectin 3)
Procedure: Long term ECG monitor — Fitting and removal of a long term ECG monitor (SpiderFlash, LivaNova)
Procedure: Monitoring ECG — Recording of automatic ECG monitor results (CSM Philips IntelliVue MP50 system)

SUMMARY:
The main hypothesis of this work is that an approach combining clinical parameters and biomarker assays could improve the understanding and prediction of the occurrence of silent atrial fibrillation (AF) in the acute phase after stroke. In this prospective work, the investigators will rely on the Dijon Stroke Registry, which collects extensive clinical data for each patient hospitalized for a stroke. As part of this registry, patients are seen 6 months after stroke to assess their clinical status. This clinical follow-up will allow us to judge the evolution of the AF diagnosed during the acute episode at a distance.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had an ischemic stroke defined according to WHO criteria and hospitalized in the Stroke Unit at the Dijon University Hospital.
* Patient 18 years of age and older
* Patient who has given oral consent

Exclusion Criteria:

* Person not affiliated to a national health insurance scheme
* Protected adult
* Pregnant or breastfeeding woman
* Patient refusing to participate in the study
* Transfer planned after the stay in the Stroke Unit to a department outside the Dijon University Hospital, not allowing for the long term screening with an external ECG monitor
* History of atrial fibrillation or atrial flutter
* Patient wearing a pacemaker or defibrillator with an atrial lead

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Diagnosis of atrial fibrillation during continuous monitoring in a Stroke unit within six months of stroke. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Didier R, Garnier L, Duloquin G, Meloux A, Sagnard A, Graber M, Dogon G, Benali K, Pommier T, Laurent G, Vergely C, Bejot Y, Guenancia C. Distribution of atrial cardiomyopathy markers and association with atrial fibrillation detected after ischaemic stroke in the SAFAS study. Stroke Vasc Neurol. 2024 Apr 30;9(2):165-173. doi: 10.1136/svn-2023-002447. PMID 37429637
- [Derived] Garnier L, Duloquin G, Meloux A, Benali K, Sagnard A, Graber M, Dogon G, Didier R, Pommier T, Vergely C, Bejot Y, Guenancia C. Multimodal Approach for the Prediction of Atrial Fibrillation Detected After Stroke: SAFAS Study. Front Cardiovasc Med. 2022 Jul 13;9:949213. doi: 10.3389/fcvm.2022.949213. eCollection 2022. PMID 35911547